CLINICAL TRIAL: NCT07184515
Title: Microbiological Study in Neck Space Infections: A Clinical and Microbiological Correlation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Hussein Abdelfatah Musa, Microbiological Study in Neck Space Infections: A Clinical and Microbiological Correlation, Assiut University
Other Study IDs: Neck space infections
Record Dates: First submitted 2025-09-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Neck Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analyze the microbiological spectrum of neck space infections and correlate it with clinical outcomes, with the goal of improving diagnostic and therapeutic approaches to these potentially serious infections & to assess the antibiotic sensitivity and resistance patterns of the isolates.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed clinically and radiologically with neck space infections.

Exclusion Criteria:

- Inadequate sample collection.

- Patients with systemic infections not originating in the neck.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed clinically and radiologically with neck space infections
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To correlate microbiological findings with clinical outcomes, including duration of hospital stay, complications, and response to therapy. | Baseline

IPD SHARING:
Plan to Share IPD: No